CLINICAL TRIAL: NCT04548102
Title: Effects of Fetal Movement Counting on Maternal and Fetal Outcome Among High Risk Pregnant Woman: A Randomized Controlled Trial
Brief Title: Effects of Fetal Movement Counting on Maternal and Fetal Outcome Among High Risk Pregnant Woman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mahmoud Abdel Ghani, Assisstant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0003381
Record Dates: First submitted 2020-08-26; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: High Risk; Pregnancy
Keywords: Fetal Movement; Maternal Outcome; Risk Pregnancy

STUDY DESIGN:
Intervention Model Description: Intervention group versus control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fetal Movement Counting (Experimental): Fetal movement counting
  Interventions: Other: Fetal movement count
- standard antenatal follow up care (No Intervention): Women in the control group received the antenatal hospital standard care.

INTERVENTIONS:
Other: Fetal movement count — Pregnant women in the study group received verbal information regarding normal fetal movements (i.e. description of the changing pattern of movement as the fetus develops, normal sleep/wake cycles, and factors which may modify the mother's perception of movements such as maternal weight and placental position), and its importance to be followed during the third trimester. A chart for fetal movements counting provided and to ensure proper performance of this task, women telephoned once a week. They also asked to show the fetal movements chart to the researcher and the health care providers in each visit. Women followed according to her antenatal visits schedule till delivery.
  Arms: Fetal Movement Counting

SUMMARY:
Up till now, there is insufficient evidence that daily fetal movement counting for pregnant women who are already have a history of high risk pregnancy is beneficial or not in term of early detection and preventing adverse pregnancy outcomes.

Aim The aim of the current study is to evaluate the effect of fetal movement counting on maternal and fetal outcome

DETAILED DESCRIPTION:
The researchers met the pregnant women in antenatal clinics during their routine follow up. Woman who was eligible to be recruited in the study signed the consent after description of the study's purpose. Pregnant women in the study group received verbal information regarding normal fetal movements (i.e. description of the changing pattern of movement as the fetus develops, normal sleep/wake cycles, and factors which may modify the mother's perception of movements such as maternal weight and placental position), and its importance to be followed during the third trimester. Further, each pregnant woman in the study group was trained how to count the fetal movement (i.e.lying down on her left side after taking her meal, and concentrating on fetal movements, calculate it three times per day, half an hour/ one time and record it in the chart). As a rule, if there are less than 10 movements felt in 2 hours, women should contact her health care provider immediately (Royal college of obstetrician & gynecologists, 2011). Fetal movements counting chart was provided and women telephoned once a week in order to ensure proper recording. They also asked to present the fetal movements' chart to the researcher and thier health care providers in each antenatal follow up visit. Pregnant women in both groups; the study and the control groups followed according to thier antenatal visits schedule till delivery. Women in the control group received the antenatal hospital standard care. The maternal and neonatal outcomes had been assessed at delivery unit.

ELIGIBILITY:
Inclusion Criteria:

* Second gravida
* Singleton
* 28 weeks gestation
* History of pregnancy induced hypertension (PIH)
* History of premature rupture of membrane (PROM)
* History of preterm labor
* History of gestational diabetes
* History of antepartum hemorrhage
* History of stillbirth
* History of fetal growth restriction

Exclusion Criteria:

* History of psychological problems
* Drugs abuse
* Experience any terrible life events during the past 6 months
* Oligohydramnios
* Multi-fetal pregnancy
* Fetal abnormalities
* Smoking

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 100 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Decreased fetal movement count | 37 weeks gestation
  Mothers' self report
Intrauterine fetal death | 37 weeks gestation
  Antenatal follow up and examination
Still birth | Within 24 hoursafter delivery
  Deliver died fetus or died within 24hrs. after delivery
NICU admission | 10 minutes after delivery
  Newborn Apgar at fifth minutes less than 6

SECONDARY OUTCOMES:
Pregnancy complications | 37 weeks gestation
  Any progress in mothers' medical conditions that affect thier pregnancy outcomes
Delivery outcome | Immediatly after delivery
  Mode of delivery and delivery complications

CONTACTS AND LOCATIONS:
Overall Officials: Rania Mahmoud A Ghani, PhD, Principal Investigator — Faculty of Nursing-Cairo University
Locations (1):
- Rania Mahmoud Abdel Ghani, Faisal, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No